CLINICAL TRIAL: NCT01784133
Title: A Phase 2, Randomized, Vehicle-Controlled, Double-Blind, Multicenter Study to Evaluate the Safety and Efficacy of Three Once-Daily CLS001 Topical Gels Versus Vehicle Administered for 12 Weeks to Subjects With Papulopustular Rosacea
Brief Title: A Twelve Week Safety and Efficacy Study in Rosacea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maruho Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLS001-CO-PR-001
Record Dates: First submitted 2013-02-01; First posted 2013-02-05 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Papulopustular Rosacea
Keywords: rosacea
MeSH Terms: conditions — Rosacea | interventions — Omiganan

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- omiganan mid dose (Active Comparator): omiganan mid dose once daily application for 12 weeks
  Interventions: Drug: omiganan
- omiganan high dose (Active Comparator): omiganan high dose once daily application for 12 weeks
  Interventions: Drug: omiganan
- Vehicle group (Placebo Comparator): Vehicle once daily application for 12 weeks
  Interventions: Drug: placebo
- omiganan low dose (Active Comparator): omiganan low dose once daily application for 12 weeks
  Interventions: Drug: omiganan

INTERVENTIONS:
Drug: omiganan
  Arms: omiganan high dose; omiganan low dose; omiganan mid dose
Drug: placebo
  Arms: Vehicle group

SUMMARY:
The purpose of this study is to evaluate th safety and efficacy of one-daily topical application of CLS001 low, mid and high dose compared to vehicle gel in subjects with papulopustular rosacea.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of papulopustular rosacea (at least 15 lesions)

Exclusion Criteria:

* nodular rosacea or subtype 3
* clinically significant abnormal findings that would interfere with study objectives

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2013-03; Primary Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change in inflammatory lesion count | 0, 1, 3, 6, 9 and 12 weeks

SECONDARY OUTCOMES:
Success on IGA defined as clear or almost clear | Week 12

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Radiant Research Inc., Birmingham, Alabama
  - ATS Clinical Research, Santa Monica, California
  - The Savin Center, PC, New Haven, Connecticut
  - Skin Care Research, Inc, Boca Raton, Florida
  - Dunedin Research Specialists, Dunedin, Florida
  - North Florida Dermatology Associates, Jacksonville, Florida
  - Dawes Fretzin Clinical Research Group, Indianapolis, Indiana
  - Grekin Skin Institute, Warren, Michigan
  - Rochester General Medical Group Center for Dermatology at Linden Oaks, Rochester, New York
  - Derm Research Center of NY Inc., Stoney Brook, New York
  - Wake Resarch, Raleigh, North Carolina
  - Oregon Dermatology and Research Center, Portland, Oregon
  - TriCities Skin and Cancer, Johnson City, Tennessee
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - Progressive Clinical Research, PA, San Antonio, Texas
  - Dermatology Research Center, Salt Lake City, Utah
  - Virginia Clinical Research Inc., Norfolk, Virginia